CLINICAL TRIAL: NCT04799301
Title: Developing Biomarkers of Dietary Intake: Dose Dependent Measurement of Sugar Intake
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 10000043; 000043-DK
Record Dates: First submitted 2021-03-13; First posted 2021-03-16 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12-15

CONDITIONS: Diet Therapy; Healthy Volunteers
Keywords: Biomarkers; Stable Isotopes; Dietary Intake
MeSH Terms: interventions — Diet

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diet with 20% of carb intake from soda (Experimental): This group will receive a weight-maintaining diet with 20% of carbohydrates provided as soda. The carbohydrates from sources other than corn and sugar cane will be reduced accordingly to meet the total carbohydrate supply.
  Interventions: Behavioral: Diet with 20% of carb intake from soda
- Diet with 50% of carb intake from soda (Experimental): This group will receive a weight-maintaining diet with 50% of carbohydrates provided as soda. The carbohydrates from sources other than corn and sugar cane will be reduced accordingly to meet the total carbohydrate supply.
  Interventions: Behavioral: Diet with 50% of carb intake from soda
- Diet with no soda (Experimental): This group will receive a weight-maintaining diet without soda. All 50% of carbohydrates will originate from sources other than corn and sugar cane.
  Interventions: Behavioral: Diet with no soda

INTERVENTIONS:
Behavioral: Diet with no soda — Weight-maintaining diet without soda, with all carbohydrates originating from sources other than corn and sugar cane
  Arms: Diet with no soda
Behavioral: Diet with 50% of carb intake from soda — Weight-maintaining diet with 50% of carbohydrates provided as soda, and all other carbohydrates originating from sources other than corn and sugar cane
  Arms: Diet with 50% of carb intake from soda
Behavioral: Diet with 20% of carb intake from soda — Weight-maintaining diet with 20% of carbohydrates provided as soda, and all other carbohydrates originating from sources other than corn and sugar cane
  Arms: Diet with 20% of carb intake from soda

SUMMARY:
Background:

Diet is one of the most modifiable behaviors affecting health. But diet assessment measures that are based on self-report can be inaccurate. Researchers want better ways to address the role of diet in chronic disease. They want to see if stable isotopes can be used to better assess what people eat.

Objective:

To see if stable isotopes can help scientists identify things people eat.

Eligibility:

Healthy adults ages 18 to 65

Design:

Participants will be screened with a medical history and physical exam. They will have blood and urine tests. These tests will be repeated during the study.

Participants will stay in the inpatient unit of the NIH in Phoenix, Arizona, for 13 weeks.

For 7 days, participants will eat a diet prepared by the NIH kitchen. They will get balanced meals that are 50% carbohydrates, 20% protein, and 30% fat. Then participants will be randomly placed on one of 3 diets containing different percentages of carbohydrates from soda.

Participants height and weight will be measured. The amount of fat and muscle in their body will be measured by body scans that are similar to x-rays.

Participants will have oral glucose tolerance tests. They will consume a sugar drink and then give blood samples over 3 hours.

Participants will give hair and stool samples.

Participants will complete a diet questionnaire. It assesses their food intake over 24 hours.

Participants will complete behavioral questionnaires and computer performance tests.

Participants will have fat biopsies taken from their stomach and thigh.

Participants will have three 24-hour stays in a metabolic chamber. It is used to measure metabolism.

DETAILED DESCRIPTION:
Study Description:

This study will be an inpatient study in which highly specific diets will be fed to volunteers for approximately 12 weeks and stable isotopes will be measured in blood, hair, and adipose. Ultimately, the goal is to develop biomarkers to be used to validate food intake patterns in outpatient clinical and epidemiological studies.

Objectives:

The primary objective of this study is to validate the use of stable isotope biomarkers as representatives of specific dietary intake patterns.

Secondary objectives include evaluation of the effect of the amount of soda on urinary sucrose and fructose excretion, extracellular vesicles levels and content, and gut microbiota.

Endpoints (Outcomes):

Primary Endpoints: Primary Endpoints: Changes in the blood, hair, and adipose carbon (13C/12C) and nitrogen (15N/14N) stable isotope ratio from baseline to 12 weeks.

Secondary Endpoints: Changes in urinary sucrose and fructose excretion, extracellular vesicles levels and content, gut microbiota from baseline to 12 weeks.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Body mass index less than or equal to 35 kg/m^2 to minimize the impact of body size on isotope measurements.
* Women and men between the ages of 18-65 years will be recruited for this study
* Healthy, as determined by medical history, physical examination, and laboratory tests.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Fasting plasma glucose greater than or equal to 126 mg/dL
* Alopecia totalis or inability to grow hair (at least one inch of hair required to obtain sample)
* Use of medication affecting metabolism and appetite in the last three months
* Medically- or self-imposed dietary restrictions that would limit a participant s ability/willingness to consume the diet to which they are randomized
* Current pregnancy, pregnancy within the past 6 months or currently lactating
* History or clinical manifestations of acute or chronic disorders or conditions that may affect appetite or EE, (such as, but not limited to type 1 or type 2 diabetes, Cushing s disease, thyroid disorders, coccidiomycoses)
* Gastrointestinal disease, including inflammatory bowel diseases (e.g. Chron s disease and ulcerative colitis), malabsorption syndromes (e.g. celiac disease), gastric ulcer (active) which may alter metabolism or absorption of study food
* Current, unstable medical conditions such as hepatitis, renal insufficiency, cancer requiring treatment in the last 5 years (except for nonmelanoma skin cancers or cancers that have clearly been cured), or central nervous system disorders etc. as assessed by history and physical exam
* Diagnosis of binge eating disorder, anorexia-nervosa, or bulimia-nervosa
* Evidence of alcohol abuse as defined by greater than or equal to 8-point score on the Alcohol consumption screening AUDIT questionnaire in adults
* Current use of tobacco products that exceed Low Dependence on the Fagerstrom Test for Nicotine Dependence Tool (score greater than 2)
* Current use of drugs such as amphetamines, cocaine, or heroin
* Any condition not specifically mentioned above that, in the opinion of the investigator, may interfere with the study or prove unsafe for participation.
* Weight change of plus or minus 5% in the last 3 months, per self report.
* Non-English speaking
* Inability of participant to understand and the unwillingness to sign a written informed consent document.

Conditions not specifically mentioned above may serve as criteria for exclusion at the discretion of the investigators. Additionally, potential subjects might be excluded if they demonstrate a style of interpersonal relationships that would inhibit successful completion of the study.

Non-English-speaking subjects as a population will be excluded from participation in this protocol. One of the secondary hypotheses of the protocol relates to a battery of psychological questionnaires and performances tests which are administered to the volunteers at the beginning and end of the study. There are currently no validated, translated forms of these questionnaires and tests available; therefore, we will restrict enrollment to English speaking subjects only.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in the blood carbon stable isotope ratio (13C/12C) from baseline to 12 weeks. | Baseline, Week 8, Week 10, Week 12
  We will test biomarker diet relationships at the week 8, 10 and 12 sampling time points, using linear mixed effects models to evaluate single CIR biomarkers of SSB in plasma. Specifically, we will also test the time x group interaction by including it as a fixed effect in the mixed model analysis to evaluate the differences in the rate of CIR change over time across groups. Baseline CIR will be included as covariate in the mixed model analysis.
Change in the hair carbon stable isotope ratio (13C/12C) from baseline to 12 weeks. | Baseline, Week 12
  We will test biomarker diet relationships at baseline and 12 weeks to determine differences in values over time and dose.

SECONDARY OUTCOMES:
Change in the carbon stable isotope ratio of alanine from baseline to 12 weeks. | Baseline, every two weeks through Week 12
  We will examine the time response of CIR-alanine. We will use a difference of 1.5 (Infinite) (+/-) from baseline as a preliminary criterion and adjust to ensure balanced representation of treatments in the 'time response' subset of participants. From these participants we will measure CIR-alanine at all timepoints. We will assess temporal change in CIR- alanine by examining week-to-week correlations to identify the time point at which biomarker measurements become independent of baseline, and by using linear mixed models to model the longitudinal trends over time.
Change in urinary sucrose/fructose over time and with varying levels of SSB intake. | Baseline, every two weeks through Week 12
  Repeated measures two-way ANOVA will be employed to assess the between-subjects effect and to compare the daily sugars excretion during different levels of sugars intake.
24h EE and its components from the metabolic chamber. | Baseline, Week 1, Week 12
  Diet-induced changes in EE will be assessed for significance using a paired t test (before/after intervention) and ANCOVA (dose).
To determine the effect of dietary changes on the microbiome of the gut, single stool samples will be collected upon admission and completion. | Baseline, Week 12
  We will measure 16s rRNA on stool samples before and after dietary intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne M Votruba, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000043-DK.html